CLINICAL TRIAL: NCT01005316
Title: Alloantibodies in Pediatric Heart Transplantation
Status: Terminated | Type: Observational
Why Stopped: Inability to meet accrual goals within the funding period.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT CTOTC-04; 7U01AI077867-02 (NIH)
Record Dates: First submitted 2009-10-27; First posted 2009-10-30 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-03

CONDITIONS: Pediatric Heart Transplantation; Pediatric Heart Transplant Recipients
Keywords: cohort study; allo-antibodies; allosensitization
MeSH Terms: interventions — Neoadjuvant Therapy; Tacrolimus; Mycophenolic Acid; Blood Component Removal; Plasmapheresis; Immunoglobulins, Intravenous; Prednisone; Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collection and biopsy tissue samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cohort A: Non-Sensitized: Cohort A will include participants who are alloantibody Luminex(TM) LABScreen. There is no study mandated care or treatment. All care given is clinical site standard of care. All sites follow a similar standard of care regimen. Non-sensitized recipients receive steroid-free maintenance immunosuppression:
  1. Induction Therapy (anti-T cell antibody induction)
  2. Tacrolimus (Prograf®)
  3. Mycophenolate Mofetil- MMF (CellCept®).
  Interventions: Drug: Induction Therapy; Drug: Tacrolimus; Drug: Mycophenolate Mofetil
- Cohort B: Sensitized: Cohort B will include participants who are alloantibody positive (Sensitized) as determined by Luminex LabScreen for Class I or Class II with specificities identified by single antigen testing.
  There is no study mandated care or treatment. All care given is clinical site standard of care. All sites follow a similar standard of care regimen.
  Sensitized recipients receive:
  1. Induction Therapy (anti-T cell antibody induction)
  2. Intraoperative plasma exchange/pheresis
  3. Short-term post-operative plasmapheresis
  4. Post-transplant course of intravenous immunoglobulin (IVIG) therapy
  5. Maintenance corticosteroids (Prednisone)
  6. Tacrolimus (Prograf®)
  7. Mycophenolate Mofetil-MMF (CellCept®).
  Interventions: Drug: Induction Therapy; Drug: Tacrolimus; Drug: Mycophenolate Mofetil; Procedure: Intraoperative plasma exchange/pheresis; Procedure: Short-term post-operative plasmapheresis; Drug: Immunoglobulins, Intravenous; Drug: Prednisone

INTERVENTIONS:
Drug: Induction Therapy — Per standard of care guidelines for immunosuppression at each clinical site.
  Other Names: anti-T cell antibody induction
Drug: Tacrolimus — Per standard of care guidelines for immunosuppression at each clinical site.
  Other Names: Prograf®
Drug: Mycophenolate Mofetil — Per standard of care guidelines for immunosuppression at each clinical site.
  Other Names: CellCept®; MMF
Procedure: Intraoperative plasma exchange/pheresis — Per standard of care guidelines for immunosuppression at each clinical site.
  Other Names: plasmapheresis
  Groups: Cohort B: Sensitized
Procedure: Short-term post-operative plasmapheresis — Per standard of care guidelines for immunosuppression at each clinical site.
  Other Names: pheresis
  Groups: Cohort B: Sensitized
Drug: Immunoglobulins, Intravenous — Post-transplant course of intravenous immunoglobulin therapy per standard of care guidelines for immunosuppression at each clinical site.
  Other Names: IVIG
  Groups: Cohort B: Sensitized
Drug: Prednisone — Maintenance corticosteroids per standard of care guidelines for immunosuppression at each clinical site.
  Other Names: corticosteroid
  Groups: Cohort B: Sensitized

SUMMARY:
The purpose of this study is to determine the clinical outcomes of sensitized pediatric heart transplant recipients with a positive donor-specific cytotoxicity crossmatch and to compare this group with outcomes in nonsensitized heart transplant recipients.

DETAILED DESCRIPTION:
There is currently a renewed interest in alloantibodies in transplantation. In 1966, Kissmeyer and colleagues reported that pre-existing antibodies directed against donor cells could cause hyperacute rejection of the renal allograft. Three years later, in a landmark study, Patel and Terasaki showed that a lymphocytotoxic assay to identify donor-specific antibodies was highly predictive of acute graft failure. These observations led to the practice of performing prospective, donor-specific crossmatches by lymphocytotoxicity assay for all kidney transplants and for heart and lung transplants when the candidate has a positive panel reactive antibody (PRA) assay. A concept evolved that transplantations should not be performed across a positive cytotoxicity crossmatch. The purpose of this study is to determine the clinical outcomes of sensitized pediatric heart transplant recipients with a positive donor-specific cytotoxicity crossmatch and to compare this group with outcomes in nonsensitized heart transplant recipients.

This study plans to enroll 370 pediatric heart transplant recipients over a period of 3 years. The follow-up period will last up to 3 years. All participants will be enrolled pretransplant. In the pretransplant phase, visits will occur every 6 months. These routine visits will continue until transplant or the end of the study. They will coincide with routine pretransplant status visits. At the time of transplant, the participants will be assigned to one of two groups. Group A will include participants who are allo-antibody negative (less than 10% by AHG CDC-PRA and ELISA in all DTT-treated serum samples). Cohort B will include participants who have the presence of a DTT-treated AHG CDC-PRA of greater than or equal to 10% and/or an ELISA-PRA greater than or equal to 10% in any pretransplant sample.

Both cohorts will receive standard transplantation care. This study has no interventions. All participants will undergo regular blood tests, and, those in the sensitized group will have additional blood testing performed after the transplant and lasting until the end of the study. Post-transplant visits will occur while participants are recovering in the hospital; at Months 1, 3, and 6; and annually until the study closes.

The information collected for the study include data from a physical exam, routine testing, adverse (AEs) and serious adverse (SAEs) events assessments, and blood collection. Each time a biopsy is done, the study will ask to review the biopsy tissue and to collect a sample. If stored tissue is not available, none will be collected.

ELIGIBILITY:
Inclusion Criteria:

* All participants listed for heart transplantation at participating CTOT-C study sites.

Exclusion Criteria:

* Listed for multiple organ transplant
* Inability or unwillingness of the participant or parent/guardian to give written informed consent or comply with the study protocol
* Condition or characteristic which in the opinion of the investigator makes the participant unlikely to complete at least one year of follow-up
* Current participation in other research studies that would, or might, interfere with the scientific integrity or safety of current study (e.g. by interference with immunosuppression management guidelines, study endpoints, excessive blood draws or SAE evaluation).

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric heart transplantation candidates
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2010-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A. Webber, MBChB, MRCP, Study Chair — University of Pittsburgh
Locations (8):
- United States (7):
  - Children's Hospital Boston, Harvard Medical School, Boston, Massachusetts
  - St. Louis Children's Hospital, Washington University, St Louis, Missouri
  - Children's Hospital of New York, Columbia University Medical Center, New York, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Children's Hospital of Philadelphia, University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
- Hospital for Sick Children, Labatt Family Heart Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Rose ML, Smith JD. Clinical relevance of complement-fixing antibodies in cardiac transplantation. Hum Immunol. 2009 Aug;70(8):605-9. doi: 10.1016/j.humimm.2009.04.016. Epub 2009 Apr 16. PMID 19375471
- [Background] Patel R, Terasaki PI. Significance of the positive crossmatch test in kidney transplantation. N Engl J Med. 1969 Apr 3;280(14):735-9. doi: 10.1056/NEJM196904032801401. No abstract available. PMID 4886455
- [Derived] Lamour JM, Mason KL, Hsu DT, Feingold B, Blume ED, Canter CE, Dipchand AI, Shaddy RE, Mahle WT, Zuckerman WA, Bentlejewski C, Armstrong BD, Morrison Y, Diop H, Ikle DN, Odim J, Zeevi A, Webber SA; CTOTC-04 investigators. Early outcomes for low-risk pediatric heart transplant recipients and steroid avoidance: A multicenter cohort study (Clinical Trials in Organ Transplantation in Children - CTOTC-04). J Heart Lung Transplant. 2019 Sep;38(9):972-981. doi: 10.1016/j.healun.2019.06.006. Epub 2019 Jun 20. PMID 31324444
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: National Heart Lung and Blood Institute (NHLBI) website — http://www.nhlbi.nih.gov/
- See also: Clinical Trials in Organ Transplantation in Children (CTOT-C) website — https://www.ctotc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrolled, Not Transplanted: These participants were consented and enrolled into the study, but did not receive a heart transplant as specified by the protocol.
- Cohort A: Non-Sensitized: Participants were enrolled into the study and received a heart transplant. Immediately prior to transplant, these participants were alloantibody negative as determined by Luminex(TM) LABScreen. All administered care was clinical site standard of care. All sites followed a similar standard of care regimen. Non-sensitized recipients received steroid-free maintenance immunosuppression: induction therapy (anti-T cell antibody induction), tacrolimus (Prograf(R)), and Mycophenolate Mofetil- MMF (CellCept(R)).
- Cohort B: Sensitized, Crossmatch Positive: Participants were enrolled into the study and received a heart transplant. Immediately prior to transplant, these participants were alloantibody positive as determined by Luminex(TM) LabScreen for Class I or Class II with specificities identified by single antigen testing. Retrospective cytotoxicity donor-specific crossmatch during their transplant procedure indicated crossmatch positivity. All administered care was clinical site standard of care. All sites followed a similar standard of care regimen. Sensitized recipients received: induction therapy (anti-T cell antibody induction), intraoperative plasma exchange/-pheresis, short-term post-operative plasmapheresis, a post-transplant course of intravenous immunoglobulin (IVIG) therapy, maintenance corticosteroids (Prednisone), tacrolimus (Prograf(R)), and Mycophenolate Mofetil- MMF (CellCept(R)).
- Cohort B: Sensitized, Crossmatch Negative: Participants were enrolled into the study and received a heart transplant. Immediately prior to transplant, these participants were alloantibody positive as determined by Luminex(TM) LabScreen for Class I or Class II with specificities identified by single antigen testing. Retrospective cytotoxicity donor-specific crossmatch during their transplant procedure indicated crossmatch negativity. All administered care was clinical site standard of care. All sites followed a similar standard of care regimen. Sensitized recipients received: induction therapy (anti-T cell antibody induction), intraoperative plasma exchange/-pheresis, short-term post-operative plasmapheresis, post-transplant course of intravenous immunoglobulin (IVIG) therapy, maintenance corticosteroids (Prednisone), tacrolimus (Prograf(R)), and Mycophenolate Mofetil- MMF (CellCept(R)).
Period: Overall Study
Arm/Group | Enrolled, Not Transplanted | Cohort A: Non-Sensitized | Cohort B: Sensitized, Crossmatch Positive | Cohort B: Sensitized, Crossmatch Negative
Started | 50 | 97 | 16 | 127
Completed | 0 | 21 | 5 | 19
Not Completed | 50 | 76 | 11 | 108
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Death | 20 | 5 | 1 | 15
Not completed — Study Termination | 5 | 63 | 9 | 85
Not completed — Lost to Follow-up | 1 | 3 | 0 | 2
Not completed — Physician Decision | 6 | 0 | 0 | 0
Not completed — Sponsor Decision | 6 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 2
Not completed — Consented to Another Study | 2 | 0 | 0 | 0
Not completed — Delisted | 8 | 0 | 0 | 0
Not completed — Transferred Care | 1 | 0 | 1 | 3
Not completed — Retransplanted | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Transplanted Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Non-Sensitized | Cohort B: Sensitized, Crossmatch Positive | Cohort B: Sensitized, Crossmatch Negative | Total
Number analyzed (Participants) | 97 | 16 | 127 | 240
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 93 | 16 | 124 | 233
  Between 18 and 65 years | 4 | 0 | 3 | 7
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.9 (6.8) | 7.8 (6.7) | 7.4 (6.3) | 7.2 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 5 | 54 | 112
  Male | 44 | 11 | 73 | 128
Region of Enrollment [Number; unit: participants]
  Canada | 12 | 1 | 18 | 31
  United States | 85 | 15 | 109 | 209

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Positive for Event of Death, Graft Loss or Rejection With Hemodynamic Compromise at 12 Months Post-Transplantation
Description: This is a composite outcome of death, graft loss or rejection with hemodynamic compromise.
  Rejection was considered to be with hemodynamic compromise if the rejection event had new onset echocardiographically measured from fractional shortening <26% with ≥5% fall from last echocardiogram or the rejection event had new onset of heart failure.
Time Frame: 12 months post-transplantation
Population: Transplanted Participants
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Non-Sensitized | Cohort B: Sensitized, Crossmatch Positive | Cohort B: Sensitized, Crossmatch Negative
Number analyzed (Participants) | 97 | 16 | 127
percentage of participants | 5.2 | 12.5 | 11.8
Statistical Analysis 1: Comparison: Cohort A: Non-Sensitized vs Cohort B: Sensitized, Crossmatch Positive vs Cohort B: Sensitized, Crossmatch Negative; The p-value compares Cohort A: Non-Sensitized with Cohort B: Sensitized, Crossmatch Positive; Test type: Superiority or Other; p = 0.2580, Fisher Exact

2. Secondary Outcome: Time to Production of Post-Transplant de Novo Donor-specific Alloantibodies
Description: Time (in days) from transplant to development of de novo donor-specific alloantibodies (DSA). This measure is calculated as time from transplant until the earliest time of development of any de novo DSA. The DSA is a newly developed alloantibody that is against the donor organ. Alloantibodies are important mediators of acute and chronic rejection.
Time Frame: Transplantation to first year post transplant (up to 12 months post transplant).
Population: Transplanted Participants
Measure: Mean (Full Range); unit: Days
Arm/Group | Cohort A: Non-Sensitized | Cohort B: Sensitized, Crossmatch Positive | Cohort B: Sensitized, Crossmatch Negative
Number analyzed (Participants) | 97 | 16 | 127
Days | 28.1 [6 to 242] | 15.4 [6 to 69] | 55.1 [7 to 355]

3. Secondary Outcome: Percentage of Participants Positive for de Novo Donor-Specific Alloantibody Production in the First Year Post-Transplantation
Description: A de novo donor-specific alloantibody (DSA) is a newly developed alloantibody that is against the donor organ. This measure includes all de novo DSA (≥1000 MFI) regardless of is persistence or timing within the first year post-transplant. Alloantibodies are important mediators of acute and chronic rejection.
Time Frame: Transplantation to first year post transplant (up to 12 months post transplant).
Population: Transplanted Participants
Measure: Number; unit: percentage of participants
Groups:
- Cohort A: Non-Sensitized: Participants were enrolled into the study and received a heart transplant. Immediately prior to transplant, these participants were alloantibody negative as determined by Luminex(TM) LABScreen. All administered care was clinical site standard of care. All sites followed a similar standard of care regimen. Non-sensitized recipients received steroid-free maintenance immunosuppression: induction therapy (anti-T cell antibody induction),
Arm/Group | Cohort A: Non-Sensitized | Cohort B: Sensitized, Crossmatch Positive | Cohort B: Sensitized, Crossmatch Negative
Number analyzed (Participants) | 97 | 16 | 127
percentage of participants | 22.7 | 50.0 | 37.8

4. Secondary Outcome: Percentage of Participants- Mortality While on Transplantation Wait-List
Description: Death that occurred while on the transplantation wait-list, and thus before receiving a heart transplant.
Time Frame: Pre-transplantation
Population: Participants Enrolled, Not Transplanted
Measure: Number; unit: percentage of participants
Arm/Group | Enrolled, Not Transplanted
Number analyzed (Participants) | 51
percentage of participants | 39.2

5. Secondary Outcome: Time From Participant Listing on Organ Wait-List to Receiving Organ Transplant, Death or De-Listing
Description: Time (in days) from listing on the organ wait-list to receiving an organ transplant, death or de-listing. This measure is calculated as time from listing on the organ wait-list until the earliest time among transplantation, death and de-listing.
Time Frame: Study enrollment to transplantation
Population: Enrolled participants who died, were transplanted or de-listed.
Measure: Mean (Full Range); unit: Days
Groups:
- Enrolled: Enrolled participants who died, were transplanted or de-listed.
Arm/Group | Enrolled
Number analyzed (Participants) | 279
Days | 128.3 [0 to 1474]

6. Secondary Outcome: Percentage of Participants With the Presence of Anti-HLA IgG Antibodies by Luminex SA Testing
Description: Luminex SA testing was used to detect the presence of anti-HLA IgG Antibodies for all samples at a central laboratory.
Time Frame: Pre-transplantation
Population: Transplanted Participants
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Non-Sensitized | Cohort B: Sensitized, Crossmatch Positive | Cohort B: Sensitized, Crossmatch Negative
Number analyzed (Participants) | 97 | 16 | 127
percentage of participants | 22.7 | 81.3 | 68.5

7. Secondary Outcome: Percentage of Participants -Quantification of Anti-HLA IgG Antibodies by Luminex SA Testing
Description: Quantification of anti-HLA IgG antibodies is measured in mean fluorescence intensity (MFI). The maximum MFI for the given subject is provided.
Time Frame: Pre-transplantation
Population: Transplanted Participants
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Non-Sensitized | Cohort B: Sensitized, Crossmatch Positive | Cohort B: Sensitized, Crossmatch Negative
Number analyzed (Participants) | 97 | 16 | 127
percentage of participants
  Missing | 0 | 0 | 2.4
  None | 77.3 | 18.8 | 29.1
  MFI 1000-3999 | 20.6 | 6.3 | 29.9
  MFI 4000-7999 | 1.0 | 12.5 | 14.2
  MFI ≥8000 | 1.0 | 62.5 | 24.4

8. Secondary Outcome: Percentage of Participants With the Presence of Anti-MICA Antibodies by Luminex TM Assay
Description: Major histocompatibility complex class I chain-related gene A (MICA) is an antigen that is a potential marker of rejection. Luminex TM assay was used to detect its presence.
Time Frame: Pre-Transplantation
Population: Transplanted Participants
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Non-Sensitized | Cohort B: Sensitized, Crossmatch Positive | Cohort B: Sensitized, Crossmatch Negative
Number analyzed (Participants) | 97 | 16 | 127
percentage of participants | 8.2 | 18.8 | 11.0

9. Secondary Outcome: Percentage of Participants -Overall Participant and Graft Survival
Description: This measure looks at the participants who did not die and/or did not receive a subsequent heart transplant.
Time Frame: Transplantation to the end of study (up to 4 years post transplant).
Population: Transplanted Participants
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Non-Sensitized | Cohort B: Sensitized, Crossmatch Positive | Cohort B: Sensitized, Crossmatch Negative
Number analyzed (Participants) | 97 | 16 | 127
percentage of participants | 93.8 | 93.8 | 87.4

10. Secondary Outcome: Presence of C4d on Endomyocardial Biopsy (EMB)
Description: The biopsy of the heart stained positive for the presence of C4d, a potential marker of rejection.
Time Frame: Transplantation to the end of study (up to 4 years post transplant).
Population: Transplanted Participants
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Non-Sensitized | Cohort B: Sensitized, Crossmatch Positive | Cohort B: Sensitized, Crossmatch Negative
Number analyzed (Participants) | 97 | 16 | 127
percentage of participants | 18.6 | 62.5 | 34.6

11. Secondary Outcome: Percentage of Participants With Occurrence of Re-Hospitalization(s)
Description: Hospitalization is defined as any hospitalization lasting greater than 24 hours.
Time Frame: Transplantation to the end of study (up to 4 years post transplant).
Population: Transplanted Participants
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Non-Sensitized | Cohort B: Sensitized, Crossmatch Positive | Cohort B: Sensitized, Crossmatch Negative
Number analyzed (Participants) | 97 | 16 | 127
percentage of participants | 66.0 | 75.0 | 62.2

12. Secondary Outcome: Percentage of Participants Positive for Severe Infection(s)
Description: Severe infections are defined as a clinical illness considered likely infectious in origin that leads to hospitalization.
Time Frame: Transplantation to the end of study (up to 4 years post transplant).
Population: Transplanted Participants
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Non-Sensitized | Cohort B: Sensitized, Crossmatch Positive | Cohort B: Sensitized, Crossmatch Negative
Number analyzed (Participants) | 97 | 16 | 127
percentage of participants | 34.0 | 43.8 | 30.7

13. Secondary Outcome: Time to Diagnosis of Chronic Rejection
Description: Time (in days) to the diagnosis of chronic rejection. Chronic rejection is defined as stenosis, irregularity, or ectasia of the epicardial vessels, or severe peripheral pruning of the distal coronary artery tree. Time to diagnosis is time from transplantation until the first diagnosis of chronic rejection.
Time Frame: Transplantation to the end of study (up to 4 years post transplant).
Population: Transplanted Participants
Measure: Mean (Full Range); unit: Days
Arm/Group | Cohort A: Non-Sensitized | Cohort B: Sensitized, Crossmatch Positive | Cohort B: Sensitized, Crossmatch Negative
Number analyzed (Participants) | 97 | 16 | 127
Days | 606.8 [264 to 1079] | NA [NA to NA] — No participants in this group were diagnosed with chronic rejection | 398.9 [4 to 1096]

14. Secondary Outcome: Time to Post-Transplantation Lymphoproliferative Disorder
Description: Time (in days) post-transplant lymphoproliferative disorder (PTLD). PTLD is defined as histopathological evidence of lymphoid proliferation (nodal or extranodal) fulfilling the criteria of the revised classification of the WHO 2008 (Swerdlow 2008). Time to PTLD is time from transplantation until the diagnosis of PTLD.
Time Frame: Transplantation to the end of study (up to 4 years post transplant).
Population: Transplanted Participants. Note to provide relevant outcome measure perspective- Of the overall number of participants analyzed, the number of diagnosed PTLD cases within groups were: Cohort A: Non-Sensitized (N=1); Cohort B: Sensitized, Crossmatch Positive (N=0); and Cohort B: Sensitized, Crossmatch Negative (N=3).
Measure: Mean (Full Range); unit: Days
Arm/Group | Cohort A: Non-Sensitized | Cohort B: Sensitized, Crossmatch Positive | Cohort B: Sensitized, Crossmatch Negative
Number analyzed (Participants) | 97 | 16 | 127
Days | 910 [910 to 910] | NA [NA to NA] — No participants in this group were diagnosed with PTLD | 118.7 [92 to 151]

15. Secondary Outcome: Time to New-Onset Diabetes Mellitus
Description: Time (in days) to new-onset diabetes mellitus. New-onset diabetes mellitus is defined as the new onset of insulin dependency or the need for oral hypoglycemic agents lasting more than 30 days post-transplant. Time to new-onset diabetes is time from transplantation until the diagnosis of new-onset diabetes.
Time Frame: Transplantation to the end of study (up to 4 years post transplant).
Population: Transplanted Participants. Note to provide relevant outcome measure perspective -Of the overall number of participants analyzed, the number of new onset diabetes mellitus cases diagnosed within groups were: Cohort A: Non-Sensitized (N=1); Cohort B: Sensitized, Crossmatch Positive (N=2); and Cohort B: Sensitized, Crossmatch Negative (N=7).
Measure: Mean (Full Range); unit: Days
Arm/Group | Cohort A: Non-Sensitized | Cohort B: Sensitized, Crossmatch Positive | Cohort B: Sensitized, Crossmatch Negative
Number analyzed (Participants) | 97 | 16 | 127
Days | 73 [73 to 73] | 48 [20 to 76] | 283.4 [5 to 965]

16. Secondary Outcome: Percentage of Participants Experiencing Acute Rejection
Description: Acute rejection is defined as any one of the following types of rejection: acute cellular rejection (International Society for Heart and Lung Transplant (ISHLT)) system for grading rejection grade 2R or greater), acute refractory cellular rejection (acute cellular rejection unresponsive to two sequential courses of corticosteroids), acute antibody mediated rejection (histological evidence of unequivocal acute capillary injury, with complement deposition and margination of macrophages with or without neutrophils), acute mixed rejection (evidence of acute antibody mediated rejection with ISHLT grade 1R or greater), or acute clinical rejection (clinically-based acute rejection, no matter the ISHLT grade, leading to an acute augmentation of immunosuppression).
Time Frame: Transplantation to the end of study.
Population: Transplanted Participants
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Non-Sensitized | Cohort B: Sensitized, Crossmatch Positive | Cohort B: Sensitized, Crossmatch Negative
Number analyzed (Participants) | 97 | 16 | 127
percentage of participants | 27.8 | 75.0 | 49.6

17. Secondary Outcome: Time to Acute Rejection
Description: Time (in days) to acute rejection. Acute rejection is defined as any one of the following types of rejection: acute cellular rejection (International Society for Heart and Lung Transplant (ISHLT) system for grading rejection grade 2R or greater), acute refractory cellular rejection (acute cellular rejection unresponsive to two sequential courses of corticosteroids), acute antibody mediated rejection (histological evidence of unequivocal acute capillary injury, with complement deposition and margination of macrophages with or without neutrophils), acute mixed rejection (evidence of acute antibody mediated rejection with ISHLT grade 1R or greater), or acute clinical rejection (clinically-based acute rejection, no matter the ISHLT grade, leading to an acute augmentation of immunosuppression). Time to acute rejection is time from transplantation to first acute rejection date.
Time Frame: Transplantation to the end of study.
Population: Transplanted Participants
Measure: Mean (Full Range); unit: Days
Arm/Group | Cohort A: Non-Sensitized | Cohort B: Sensitized, Crossmatch Positive | Cohort B: Sensitized, Crossmatch Negative
Number analyzed (Participants) | 97 | 16 | 127
Days | 151.0 [8 to 991] | 74.5 [6 to 608] | 124.7 [4 to 933]

ADVERSE EVENTS:
Time Frame: Transplantation through end of study (up to 3 years)
Description: Only serious adverse events were collected.
Arm/Group | Cohort A: Non-Sensitized | Cohort B: Sensitized, Crossmatch Positive | Cohort B: Sensitized, Crossmatch Negative
All-Cause Mortality (participants affected / at risk) | 5/97 | 1/16 | 16/127
Serious Adverse Events (participants affected / at risk) | 30/97 | 7/16 | 43/127
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Non-Sensitized (N=97) | Cohort B: Sensitized, Crossmatch Positive (N=16) | Cohort B: Sensitized, Crossmatch Negative (N=127)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure high output (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial reperfusion injury (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Torsade de pointes (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Serum sickness (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Transplant rejection (Immune system disorders) | 0 (0) | 2 (2) | 5 (6)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 2 (3)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungal endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 4 (4) | 0 (0) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Neutropenic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Graft dysfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Transplant failure (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Epstein-Barr virus associated lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary vein stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Arterial thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study enrollment closed December 2013:target enrollment was not met (78% of target).Not all participants recv'd the planned 3 year follow-up. Participants were followed for a year after enrollment closure then enrolled into CTOTC-09 (NCT02752789).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No